CLINICAL TRIAL: NCT05149209
Title: One-Year Clinical Evaluation of a Fluoride, Calcium and Phosphate-Releasing New Bioactive Material Versus a Fluoride-Releasing Hybrid Restorative Material in Cervical Lesions: A Randomized Clinical Trial.
Brief Title: Evaluation of a New Bioactive Material Versus a Fluoride-Releasing Hybrid Restorative Material in Cervical Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Khaled Mohamed Samir, Resident at Conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: cons2021
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Controlled Trial. Trial type: Two, Parallel arm design. Trial framework: Equivalence frame Allocation ratio: 1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will be blinded to the technique used since the patient will attend the same number of visits and he can not differentiate between different restorative materials.
  The operator cannot be blinded because of the difference in the application procedures of each restorative material.
  The outcome assessor will be blinded to the material used. This will be performed by M.S. and Y.H. Therefore the assessors mustn't be included in the preclinical assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride, calcium and phosphate-releasing new bioactive material (Activa™ Presto, Pulpdent®, USA). (Experimental): ACTIVA Presto is a novel bioactive material with a mineral-enriched hydrophilic resin base and a patented rubberized component that resists abrasion and wear with high release and recharge of not only fluoride but also calcium and phosphate ions. It doesn't contain BIS-GMA, Bisphenol A, or BPA derivatives.
  Interventions: Procedure: cervical restoration
- Fluoride-releasing hybrid restorative material (Giomer, Shofu, Japan). (Active Comparator): Giomer is a hybrid restorative material that contains a resin base and pre-reacted glass ionomer. S-PRG (surface reaction type) technology provides some properties of GI such as fluoride release and recharge which helps prevent recurrent caries.
  Interventions: Procedure: cervical restoration

INTERVENTIONS:
Procedure: cervical restoration — A class v cavity will be prepared after local anesthesia has been given as required. Rubber dam isolation will be done. Selective enamel etching and a universal adhesive agent (Beautibond, Shofu, Japan) will be applied over all the cavity surfaces. Followed by, placement of restorative material according to the randomization sequence. Finally, restoration finishing and polishing will be done.

SUMMARY:
* This study will be conducted to evaluate and compare the clinical performance of fluoride, calcium, and phosphate-releasing new bioactive material versus a fluoride-releasing hybrid restorative material in cervical lesions for one-year follow-up.
* The clinical evaluation will be done using modified USPHS criteria at baseline,3,6,9 and 12 months.

DETAILED DESCRIPTION:
two groups of 30 patients will receive cervical restorations by using calcium and phosphate releasing hybrid restorative material (Activa™ Presto, Pulpdent®, USA), or a fluoride-releasing hybrid restorative material (Giomer, Shofu, Japan). Then these restorations will be evaluated at baseline, 3 months, 6 months, 9 months, and 12 months according to modified USPHS criteria in terms of marginal adaptation, Marginal discoloration, recurrent caries, retention, surface texture, and Post-operative sensitivity.

* Examination and selection of all patients will be done according to inclusion and exclusion criteria.
* A class v cavity will be prepared after local anesthesia has been given as required. Rubber dam isolation followed by the placement of restorative material according to the randomization sequence.
* For the intervention: selective etching to enamel and universal bond agent to all the cavity will be applied first, followed by filling of the cavity with fluoride, calcium, and phosphate-releasing new bioactive material (Activa™ Presto, Pulpdent®, USA) using a 19-gauge applicator tip on the syringe and light-curing for 20 seconds between each 2mm layer.
* For the control group: selective etching to enamel and universal bond agent to all the cavity will be applied first, followed by filling of the cavity with fluoride-releasing hybrid restorative material (Giomer, Shofu, Japan) and will be light polymerized using a light-emitting diode (LED) light-curing unit for 10 seconds between each 2mm layer.

ELIGIBILITY:
Inclusion Criteria:

* a)Inclusion Criteria of participants:

  * Male or female gender.
  * Only co-operative patients will be approved to participate in the trial.
  * Medically free adult patients.
  * The age range of the patients is 18-40 years. b)Inclusion Criteria of teeth:
  * Small to moderate cervical lesion.
  * Vital upper or lower teeth with no signs of irreversible pulpitis.
  * Caries extension shouldn't exceed mesiodistal width and inciso(occluso)-gingival length not exceed incisal (occlusal) one third.

Exclusion Criteria:

* a)Exclusion criteria of participants:

  * Allergic history concerning methacrylates
  * Pregnancy
  * Heavy smoking; xerostomia
  * Lack of compliance
  * Patients with disabilities.
  * Patients having systemic diseases or severe medically compromised.
  * Patients with severe bruxism, clenching, or temporomandibular joint disorders.

    b)Exclusion criteria of the teeth:
  * Deep defects (close to the pulp, less than 1 mm distance).
  * Periapical pathology or signs of pulpal pathology.
  * Possible prosthodontic restoration of teeth.
  * Heavy occlusion and occlusal contacts or history of bruxism.
  * Pulpitis, non-vital or endodontically treated teeth.
  * Sever periodontal affection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | one year
  The restoration will be clinically assessed by visual inspection and explorer. Restorations will be given a score using modified USPHS criteria:
  Alfa: Closely adapted, no visible crevice Bravo: Visible crevice, the explorer will penetrate Charlie: Crevice in which dentin is exposed

SECONDARY OUTCOMES:
Marginal Discoloration | one year
  Clinical evaluation by visual inspection and mirror if needed using modified USPHS criteria. Restorations will be given the score:
  Alfa if No discoloration Bravo if Non penetrating marginal discoloration which can be polished away Charlie if Discoloration with penetration in pulpal direction.
Retention | one year
  Clinical evaluation by visual inspection and explorer. Restorations will be given a score according to modified USPHS criteria :
  Alfa if restoration is retained and there is no loss of restoration. Charlie if loss of restoration.
Secondary caries | one year
  Clinical evaluation by visual inspection and explorer. Restorations will be given a score according to modified USPHS criteria:
  Alfa if no recurrent caries is detected, charlie if recurrent caries is detected.
  .
surface texture | one year
  Clinical evaluation by visual inspection and explorer. Restorations will be given a score according to modified USPHS criteria:
  Alfa if restoration is enamel-like surface Bravo if Surface rougher than enamel, clinically acceptable Charlie if Surface is unacceptably rough.
postoperative sensitivity | one year
  Verbal evaluation by asking the patient. Restorations will be given a score according to modified USPHS criteria:
  Alfa if not present Bravo if sensitive but diminishing in intensity Charlie if constant sensitivity not diminishing.

CONTACTS AND LOCATIONS:
Locations (1):
- Nourhan Khaled Mohamed Samir, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Yes
* Full protocol will be published online in Clinicaltrials.gov to avoid repetition, and keep the integrity of the research work.
  * Thesis will be discussed and defended in front of a judging committee.
  * The study will be published to report the results of this clinical trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 24 months
Access Criteria: open access